CLINICAL TRIAL: NCT04462601
Title: Descriptive Study of Variations in Serum Translocation Markers of the Intestinal Microbiota in Patients With Gougerot-Sjögren Syndrome According to Disease Activity
Acronym: IMISS
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: NIMAO/2019-01/RG-01
Record Dates: First submitted 2020-07-03; First posted 2020-07-08 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, blood, stool and saliva
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Sjögren Syndrome
  Interventions: Other: Biomarker detection

INTERVENTIONS:
Other: Biomarker detection — Quantification of serum markers of intestinal permeability and bacterial and fungal translocation

SUMMARY:
Gougerot-Sjögren syndrome or Sjögren syndrome is a chronic autoimmune disease belonging to connectivitis, the classic triad of symptoms being the association of a sicca syndrome (generally predominant in the mouth and / or ocular, but also present at the cutaneous, vaginal or tracheal level), diffuse arthromyalgia and marked fatigue. The study investigators hypothesize that changes in the gut microbiota, by modulating gut permeability and thereby promoting microbial translocation, would have immunomodulatory effects that could be correlated to changes in the activity of Gougerot-Sjögren disease.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be a member or beneficiary of a health insurance plan
* Patients with primary Sjögren's syndrome according to the AECG criteria

Exclusion Criteria:

* The subject is participating in a category I interventional study, or is in a period of exclusion determined by a previous study
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Pregnant, parturient or breastfeeding patients
* Patients with secondary Sjögren's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (≥ 18 years old) with primary Sjögren's syndrome according to the AECG criteria and / or validation by an expert, subject to their agreement, followed in one of the departments participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-11-13 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Difference in Intestinal Fatty Acid Binding Protein (I-FABP) levels from baseline in patients passing to a different level of disease activity | Upon changing disease activity level (maximum 3 years)
  ng/ml measured by ELISA; Change in disease activity levels defined by 3-point change on the European League Against Rheumatism Sjögren Syndrome Disease Activity Index (ESSDAI)
Difference in zonulin-1 levels from baseline in patients passing to a different level of disease activity | Upon changing disease activity level (maximum 3 years)
  ng/ml measured by ELISA; Change in disease activity levels defined by 3-point change on the European League Against Rheumatism Sjögren Syndrome Disease Activity Index (ESSDAI)

SECONDARY OUTCOMES:
Difference in LPS-binding Protein levels from baseline in patients passing to a different level of disease activity | Upon changing disease activity level (maximum 3 years)
  pg/ml, measured by ELISA; Change in disease activity levels defined by 3-point change on the European League Against Rheumatism Sjögren Syndrome Disease Activity Index (ESSDAI)
Difference in LPS-binding Protein levels from baseline in patients reporting an improvement in disease activity | Upon changing disease activity level (maximum 3 years)
  pg/ml, measured by ELISA; patient-reported disease severity defined by 1-point increase on the European League Against Rheumatism Sjögren's syndrome Patient Reported Index (ESSPRI)
Difference in LPS-binding Protein levels between patients receiving or not systemic treatment (corticosteroids, plaquenil or methotrexate) | Upon changing disease activity level (maximum 3 years)
  pg/ml, measured by ELISA
Difference in soluble CD14 levels from baseline in patients passing to a different level of disease activity | Upon changing disease activity level (maximum 3 years)
  ng/ml, measured by ELISA; Change in disease activity levels defined by 3-point change on the European League Against Rheumatism Sjögren Syndrome Disease Activity Index (ESSDAI)
Difference in soluble CD14 levels from baseline in patients reporting an improvement in disease activity | Upon changing disease activity level (maximum 3 years)
  ng/ml, measured by ELISA; patient-reported disease severity defined by 1-point increase on the European League Against Rheumatism Sjögren's syndrome Patient Reported Index (ESSPRI)
Difference in soluble CD14 levels between patients receiving or not systemic treatment (corticosteroids, plaquenil or methotrexate) | Upon changing disease activity level (maximum 3 years)
  ng/ml, measured by ELISA
Difference in fungal 18s RNA levels from baseline in patients passing to a different level of disease activity | Upon changing disease activity level (maximum 3 years)
  PCR and sequencing; Change in disease activity levels defined by 3-point change on the European League Against Rheumatism Sjögren Syndrome Disease Activity Index (ESSDAI)
Difference in fungal 18s RNA levels from baseline in patients reporting an improvement in disease activity | Upon changing disease activity level (maximum 3 years)
  PCR and sequencing; patient-reported disease severity defined by 1-point increase on the European League Against Rheumatism Sjögren's syndrome Patient Reported Index (ESSPRI)
Difference in fungal 18s RNA levels between patients receiving or not systemic treatment (corticosteroids, plaquenil or methotrexate) | Upon changing disease activity level (maximum 3 years)
  PCR and sequencing
Difference in bacterial 16s RNA levels from baseline in patients passing to a different level of disease activity | Upon changing disease activity level (maximum 3 years)
  PCR and sequencing; Change in disease activity levels defined by 3-point change on the European League Against Rheumatism Sjögren Syndrome Disease Activity Index (ESSDAI)
Difference in bacterial 16s RNA levels from baseline in patients reporting an improvement in disease activity | Upon changing disease activity level (maximum 3 years)
  PCR and sequencing; patient-reported disease severity defined by 1-point increase on the European League Against Rheumatism Sjögren's syndrome Patient Reported Index (ESSPRI)
Difference in bacterial 16s RNA levels between patients receiving or not systemic treatment (corticosteroids, plaquenil or methotrexate) | Upon changing disease activity level (maximum 3 years)
  PCR and sequencing
EQ-5D-5L questionnaire | Baseline
  score 0-100
EQ-5D-5L questionnaire | Upon changing disease activity level (maximum 3 years)
  score 0-100
World Health Organization Quality Of Life BREF questionnaire | Baseline
  score 0-100
World Health Organization Quality Of Life BREF questionnaire | Upon changing disease activity level (maximum 3 years)
  score 0-100
Hospital Anxiety and Depression Scale | Baseline
  score 0-42
Hospital Anxiety and Depression Scale | Upon changing disease activity level (maximum 3 years)
  score 0-42
Multidimensional Fatigue Inventory | Baseline
  score 4-20
Multidimensional Fatigue Inventory | Upon changing disease activity level (maximum 3 years)
  score 4-20

CONTACTS AND LOCATIONS:
Overall Officials: Radjiv Goulabchand, Principal Investigator — CHU Nimes
Locations (1):
- CHU de Nimes, Nîmes, France